CLINICAL TRIAL: NCT06804083
Title: Oral Immunoglobulins From Bovine Colostrum and Anti-inflammatory Extracts in Patients With Chronic Prostatitis/Chronic Pelvic Pain Syndrome: A Prospective Study
Brief Title: Bovine Colostrum Efficacy for the Treatment of Chronic Prostatitis Symptoms.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Clinica Urologica Molinette - Città della Saliute e della Scienza (Other)
Collaborators: A.O.U. Città della Salute e della Scienza - Molinette Hospital (Other)
Responsible Party: Principal Investigator, Mattia Sibona, Urologist, MD, Clinica Urologica Molinette - Città della Saliute e della Scienza
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CET n. 00054/2019
Record Dates: First submitted 2025-01-08; First posted 2025-01-31 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Chronic Prostatitis (CP); Chronic Prostatitis With Chronic Pelvic Pain Syndrome; Chronic Prostatitis/ Pelvic Pain Syndrome
Keywords: Chronic prostatitis; chronic pelvic pain syndrome; PROSTYM®; bovine colostrum; LUTS; pain
MeSH Terms: conditions — Prostatitis; Pain

STUDY DESIGN:
Intervention Model Description: prospective, observational, single-arm study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- PROSTYM® (Experimental): It is a phytotherapic drug. The composition of PROSTYM® (per capsule) includes bovine colostrum (30 mg), Serenoa extracts (320 mg), glutathione (30 mg), N-acetyl cysteine (20 mg), Ribes nigrum extracts (50 mg), willow extracts (50 mg), zinc (5 mg), selenium (27.5 micrograms), and vitamin E (6 mg). All these components are included in one capsule. The drug is administered for 6 months in a 1 cp/die dosage.
  Interventions: Drug: oral combination of colostrum and Serenoa repens extracts (PROSTYM®)

INTERVENTIONS:
Drug: oral combination of colostrum and Serenoa repens extracts (PROSTYM®) — The composition of PROSTYM® (per capsule) includes bovine colostrum (30 mg), Serenoa extracts (320 mg), glutathione (30 mg), N-acetyl cysteine (20 mg), Ribes nigrum extracts (50 mg), willow extracts (50 mg), zinc (5 mg), selenium (27.5 micrograms), and vitamin E (6 mg).
  Drug administration (1 capsule per day) for 6 months.
  Other Names: PROSTYM®

SUMMARY:
Chronic prostatitis/chronic pelvic pain syndrome (CP/CPPS) is a bothering condition characterized by pain localized to the pelvic, perineal and/or genital area and lower urinary tract symptoms (LUTS). Phytotherapy, which involves the combination of two or more active compounds, can be used to treat this challenging condition.

The aim of this study was to investigate the role of an oral combination of colostrum and Serenoa repens extracts (PROSTYM®) in the treatment of CP/CPPS patients. The main questions the present study aims to answer are:

* Does PROSTYM® enhance quality of life of CPP/CPPS patients?
* Does it help reducing pain symptoms of CPP/CPPS patients?

Researchers will investigate whether PROSTYM® works to treat CPP/CPPS symptoms, so its efficacy, but also its tolerability and adherence to therapy.

Participants will:

* Take PROSTYM® every day for 6 months;
* Visit the clinic for follow-up visits at 3 and 6 months;
* Answer validated questionnaires and declare potential adverse events at follow-up visits.

ELIGIBILITY:
Inclusion Criteria:

* adult male patients (aged >18 years)
* clinical affection by CP/CPPS with symptoms that persisted for ≥6 months;
* CPSI pain domain score ≥5 points;
* negative Meares and Stamey test score.

Exclusion Criteria:

* patients with prevalent BPH symptoms (CPSI pain domain <5), acute prostatitis, chronic bacterial prostatitis (positive Meares and Stamey test), prostate or bladder cancer, urethral stenosis or neurological bladder;
* no other drug or supplement specific to chronic prostatitis in the previous 30 days.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male patients (with a prostate)
Enrollment: 42 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Rate of ≥25% Decrease in CPSI Total Score Compared to Baseline | 6 months
  improvement of CP symptoms

SECONDARY OUTCOMES:
Rate of ≥25% Decrease in CPSI Pain Domain Score Compared to Baseline | 6 months
  improvement of CP pain symptoms
Rate of ≥25% Decrease in CPSI QoL Domain Score Compared to Baseline | 6 months
  improvement of CP QoL
Total Number of Adverse Events | 6 months
  number and type, so safety analysis

CONTACTS AND LOCATIONS:
Locations (1):
- Molinette Hospital, Torino, Torino, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wagenlehner FM, Schneider H, Ludwig M, Schnitker J, Brahler E, Weidner W. A pollen extract (Cernilton) in patients with inflammatory chronic prostatitis-chronic pelvic pain syndrome: a multicentre, randomised, prospective, double-blind, placebo-controlled phase 3 study. Eur Urol. 2009 Sep;56(3):544-51. doi: 10.1016/j.eururo.2009.05.046. Epub 2009 Jun 3. PMID 19524353
- [Background] Litwin MS, McNaughton-Collins M, Fowler FJ Jr, Nickel JC, Calhoun EA, Pontari MA, Alexander RB, Farrar JT, O'Leary MP. The National Institutes of Health chronic prostatitis symptom index: development and validation of a new outcome measure. Chronic Prostatitis Collaborative Research Network. J Urol. 1999 Aug;162(2):369-75. doi: 10.1016/s0022-5347(05)68562-x. PMID 10411041
- [Background] Cai T, Luciani LG, Caola I, Mondaini N, Malossini G, Lanzafame P, Mazzoli S, Bartoletti R. Effects of pollen extract in association with vitamins (DEPROX 500(R)) for pain relief in patients affected by chronic prostatitis/chronic pelvic pain syndrome: results from a pilot study. Urologia. 2013 Apr 24;80 Suppl 22:5-10. doi: 10.5301/RU.2013.10597. Epub 2013 Jan 16. PMID 23334883
- [Background] Sibona M, Destefanis P, Agnello M, Lillaz B, Giuliano M, Cai T, Gontero P. The association of Boswellia resin extract and propolis derived polyphenols can improve quality of life in patients affected by prostatitis-like symptoms. Arch Ital Urol Androl. 2020 Jan 14;91(4):251-255. doi: 10.4081/aiua.2019.4.251. PMID 31937091